CLINICAL TRIAL: NCT03290846
Title: Secretin Increases Glucose Uptake in Human Brown Adipose Tissue and Induces Satiation.
Brief Title: Secretin Activates Human Brown Fat and Induces Satiation.
Acronym: GUTBAT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Pirjo Nuutila, Professor, MD PhD, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T153/2016
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Secretin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single blinded randomised study, secretin infusion is given on one day, saline infusion on an other day.
Masking Description: Participants receive drug and placebo infusion without knowing which day is which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Secretin study (Experimental): PET and MRI scannings will be performed twice. Subjects will be given secretin hydrochloride and placebo on separate days. In addition, subjects will undergo cold exposure PET scanning once.
  Interventions: Drug: Secretin Human; Drug: Saline Solution; Other: Cold exposure

INTERVENTIONS:
Drug: Secretin Human — Randomized, single-blinded secretin hydrochloride infusion.
Drug: Saline Solution — Randomized, single-blinded saline infusion.
Other: Cold exposure — All subjects will undergo a cold exposure PET scan.

SUMMARY:
15 healthy males will be studied with PET/CT, using FDG to investigate glucose metabolism, and radiowater to investigate perfusion. One scan will be performed in controlled cold exposure, to see whether subjects have cold activated brown adipose tissue. Two scans will be performed in room temperature conditions, where all subjects are blinded and randomised to receive placebo and secretin hydrochloride. PET/CT scans will be analysed blinded.

20 healthy males will also be studied with fMRI, in order to investigate brain activity responses to appetizing versus bland foods. This study will be conduced on the same patients as the PET/CT study, but additional subjects with same inclusion and exclusion criteria will be recruited. Two fMRI scans will be performed in room temperature conditions, where all subjects are blinded and randomised to receive placebo and secretin hydrochloride. fMRI scans will be analysed blinded.

DETAILED DESCRIPTION:
The PET/CT study will consist of 15 healthy, normal weight males, between ages 18-65. A 2-hour oral glucose tolerance test is performed on screening day. Calorimetry data is collected at baseline (resting and fasting) condition.

Three PET/CT scans on three different days will be performed to all 15 study subjects. Radiowater (15O)-H2O is used to study perfusion and FDG ((F18)-FDG) to study glucose metabolism. After radiowater, PET data is collected from the neck area for 6 minutes. After FDG, PET data is collected for 40 minutes on the neck area, 15 minutes on the chest, 15 minutes on the abdomen and 15 minutes on the brain. Calorimetry is collected during the entire scan. Blood samples are collected during scans for metabolites and for a plasma activity curve.

One scan is performed during controlled, cold exposure. This is done to investigate, whether patients have cold activated brown adipose tissue. After this, subjects will undergo two room temperature condition scans on different days, where participants are single-blinded and randomised to receive placebo (saline) or secretin (secretin hydrochloride) infusions. All scans are done in fasting conditions. After subjects have fed at the PET centre, calorimetry data is collected on all days.

A full body MRI will be performed on a separate day with the Dixon-method.

After scanning visits, brown adipose tissue biopsies will be taken from volunteers by a plastic surgeon. These samples are analysed in Munich.

Dynamic scan data is analysed with the Carimas program, using Patlak plot. Analysis is performed blinded. Further statistics analysis is done with SPSS.

The fMRI study will consist of 20 healthy, normal weight males, between ages 18-65. Subjects who underwent PET/CT scanning will be recruited for this study, as well as an additional group of subjects with the same inclusion and exclusion criteria. A 2-hour oral glucose tolerance test is performed on screening day for additional subjcts.

Two fMRI scans are conducted in room temperature after overnight fast on separate days. Subjects are randomized and blinded to receive placebo and secretin hydrochloride on separate days. Data on brain activity while viewing appetizing versus bland food images is collected during scan. After scanning subjects are given a meal and then followed up for two hours. Data on subjective satiety will be collected with a visual analogue scale questionnaire on nine different timepoints during the day: in preprandial, prandial and postprandial conditions.

Functional MRI data is analyzed with Matlab. Analysis is performed blinded. Satiety score is analzed with SPSS.

ELIGIBILITY:
Inclusion Criteria:

* healthy normal weight

Exclusion Criteria:

* cardiovascular disease, diabetes
* smoking

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Radiation exposure for fertile women is avoided
Enrollment: 23 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Secretin activates brown fat | Effect within one hour
  Secretin increases brown adipose tissue glucose uptake compared to placebo. This is studied with PET/CT, using a glucose tracer.
Secretin activates brown fat | Effect within six minutes
  Secretin increases brown adipose tissue flow compared to placebo. This is studied with PET/CT, using a radiowater tracer.
Secretin induces satiation | Effect within one hour
  Secretin attenuates brain activity, when subjects are viewing palatable vs. non-palatable food images.

SECONDARY OUTCOMES:
Secretin increases whole body energy expenditure | Effect within two hours
  Secretin increases whole body energy expenditure compared to placebo. Data is collected durin PET/CT scans by indirect calorimetry.
Secretin induces satiety | Effect within three hours
  Composite satiety score is measured by visual analogue scale questionnaire
Secretin reduces food consumption. | Within three days
  Data on food consumption is collected directly after scan, as well as with food diaries. Calory intake is measured and comparisons are made between secretin and placebo.

OTHER OUTCOMES:
Secretin induces changes in biomarkers and metabolites. | Within two hours
  Serum samples are collected during PET/CT scan and analyzed.
Brown adipose tissue biopsies. | Within 2 months
  Brown adipose tissue biopsy samples are collected from subjects and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo R Nuutila, MD,PhD, Principal Investigator — Turku UH
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
No data, where participants could be identifiable, will be shared.

REFERENCES:
- [Derived] Sun L, Laurila S, Lahesmaa M, Rebelos E, Virtanen KA, Schnabl K, Klingenspor M, Nummenmaa L, Nuutila P. Secretin modulates appetite via brown adipose tissue-brain axis. Eur J Nucl Med Mol Imaging. 2023 May;50(6):1597-1606. doi: 10.1007/s00259-023-06124-4. Epub 2023 Feb 11. PMID 36764966
- [Derived] Laurila S, Rebelos E, Lahesmaa M, Sun L, Schnabl K, Peltomaa TM, Klen R, U-Din M, Honka MJ, Eskola O, Kirjavainen AK, Nummenmaa L, Klingenspor M, Virtanen KA, Nuutila P. Novel effects of the gastrointestinal hormone secretin on cardiac metabolism and renal function. Am J Physiol Endocrinol Metab. 2022 Jan 1;322(1):E54-E62. doi: 10.1152/ajpendo.00260.2021. Epub 2021 Nov 22. PMID 34806426
- [Derived] Laurila S, Sun L, Lahesmaa M, Schnabl K, Laitinen K, Klen R, Li Y, Balaz M, Wolfrum C, Steiger K, Niemi T, Taittonen M, U-Din M, Valikangas T, Elo LL, Eskola O, Kirjavainen AK, Nummenmaa L, Virtanen KA, Klingenspor M, Nuutila P. Secretin activates brown fat and induces satiation. Nat Metab. 2021 Jun;3(6):798-809. doi: 10.1038/s42255-021-00409-4. Epub 2021 Jun 21. PMID 34158656